CLINICAL TRIAL: NCT01871012
Title: The Assessment of the Management of Intraoperation and Postoperative Quality of Recovery for Total Knee Replacement in Elder Diabetic Patients
Brief Title: The Assessment of Postoperative Recovery in Elder Diabetic Patients
Acronym: TKRDM2013
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Chinese PLA General Hospital (Other)
Responsible Party: Principal Investigator, Junle Liu, Principal Investigator, Chinese PLA General Hospital
Other Study IDs: TKRPLA2013
Record Dates: First submitted 2013-06-04; First posted 2013-06-06 (Estimated); Last update posted 2013-10-16 (Estimated); Status verified 2013-10

CONDITIONS: Anesthesia; Knee Osteoarthritis
Keywords: Nerve Block; Intraoperative Care; Postoperative Recovery and Complications; Stress and Inflammation
MeSH Terms: conditions — Osteoarthritis, Knee; Inflammation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 7 Days
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- non-diabetes mellitus group: Subjects undergoing Total Knee Replacement are not diagnosed with diabetes mellitus.
- diabetes mellitus group: subjects have been diagnosed diabetes mellitus mora than three years without serious nerve system complications.

SUMMARY:
Total Knee Replacement (TKR) performed under general anesthesia is a common successful orthopedic procedure. Nonetheless, in elder patients with diabetes mellitus (DM) this procedure can present unique challenges to orthopedic surgeon and anesthesiologist alike. Many diabetic patients have clinical or subclinical neuropathy. Although there is no evidence that the neuropathy is exacerbated by neural blockade, recent studies have suggested that the peripheral nerves in diabetic patients may be more susceptible to trauma and local anaesthetic toxicity. Therefore, The investigators observe peripheral nerve blocks with ropivacaine on diabetic patients or non-diabetic patients undergoing TKR by assessing the management of intraoperation and the Postoperative Recovery and complications.

DETAILED DESCRIPTION:
After standard external monitors, pulse oximeter, electrocardiogram, noninvasive blood pressure, were applied on subject's arrival in the operation room. Subjects had an intravenous line placed in the upper extremity. Patients received midazolam (0.015-0.03 mg.kg-1), sulfentanil (0.10-0.15µg.kg-1) by infusion, in divided doses, before lumbar plexus and sciatic nerve blocking and supplemental 100% oxygen (3 L.min-1) was administered by facemask spontaneously breathing during the procedure. The procedure was performed by two anesthesiologists with extensive experience in nerve block. After sterile preparation and draping, PNBs were administered using a 21-gauge, 100-mm Stimuplex block needle and a nerve stimulator. A posterior approach to lumbar plexus block was performed with patient in the lateral decubitus position and after a quadriceps muscle response had been identified with nerve stimulator settings at 2 HZ frequency and current between 0.3 and 0.5 mA, and 0.2% ropivacaine (25-30 mL) was injected slowly. Sciatic nerve block was performed in the same position after a twitch of hamstrings, soleus, foot, or toes, had been elicited using the similar current, and 0.2% ropivacaine (15-20 mL) was injected slowly.

After nerve blocks finished, a standardized balanced anesthetic technique was provided in both groups. Anesthesia was administered with etomidate (0.1-0.2mg.kg-1) and rocuronium (0.4-0.6 mg.kg-1), and then suitable laryngeal mask airway (LMA) was facilitated with a respiratory rate of 10-12 bpm, an I:E ratio of 1:2 and an FiO2 of 0.6. Tidal volume will be adjusted to an end tidal CO2 of 35-40 mmHg. Maintaining with remifentanil (0.05-0.30 µg.kg-1.min-1), target concentrations of propofol (0.3-2.0 µg.mL-1) and sevoflurane (0.4 MAC). Infusion rates of propofol and remifentanil varied according to clinical judgment and bispectral index (BIS) range between 40 and 60. All procedures were performed by two veteran anesthesiologists.

Every patient shows signs of inadequate anesthesia such as an increase in systolic arterial blood pressure > 20% from baseline or a heart rate greater than 90 in the absence of hypovolemia, sweating, flushing or movement, sulfentanil, 5-10µg, may be administered. Persistent hypertension without signs of inadequate anesthesia will be treated with nicardipine, 0.4 mg IV, every 3 min until return to baseline value. In both groups patients with a heart rate less than 50 bpm not correlated with blood pressure variation will receive atropine 0.3 mg every 3 minutes until heart rate is back to at least 50 bpm. In all patients, from anesthetic induction to end of surgery, a decrease in systolic blood pressure of more than 30% less than baseline values will be treated with ephedrine 6 mg or phenylephrine 100 µg every 3 min until return to baseline value. Propofol will be stopped at completion of skin closure. Intraoperatively, each patient will also receive 2 mg of tropisetron to decrease postoperative nausea.

Postoperative pain was controlled for all patients routinely by intravenous sulfentanil patient-controlled analgesia (PICA) in combination with Parecoxib (40 mg, every 12 h), a selective COX-2 inhibiter. PICA was continued with sulfentanil (0.9µg.h-1) and 0.9 µg sulfentanil bolus with a 8-min lockout time. Oral oxycodone 0.2 mg was administered necessarily.

The doses of all IV drugs and duration of anesthesia and surgery will be recorded. Ephedrine and phenylephrine consumption and the amount of intravascular fluid administration and all the intraoperative drug dose adjustments will be recorded. The esophageal temperature of the patients will be monitored and maintained at 36 ℃using a force-air warming blanket and warmed i.v. fluids. Postoperative Recovery of the PQRS will be measured on presurgery, 15 minute, 40 minute, 1 day, 3day, 7day postoperatively.

Cardiovascular, cerebrovascular and Pulmonary complications (7days postoperation ), C-reacting protein (CRP) measured preoperatively and on 1, 3 and 7 day postoperatively. Erythrocyte Sedimentation Rate (ESR) measured preoperatively and on 1, 3 and 7 day postoperatively, IL-6 measured preoperatively and on 1, 3 and 7 day postoperatively;blood sugar measured preoperatively on 1, 3 and 7 day postoperatively, nervous system complications and charge measured before left hospital.

ELIGIBILITY:
Inclusion Criteria:

* Age > 65 years old;
* Undergoing selective total uni-knee replacement surgery;
* American Society of Anesthesiologists (ASA) physical status I-III;
* Mini-Mental score examination (MMSE) being more than 23;
* Diagnosis of Type 2 diabetes > 3 years or No diabetes.

Exclusion Criteria:

* Patient refusal to participate in the study;
* Patient refusal of regional block;
* Allergic to local anesthetics or general anesthetics;
* History of opioid dependence;
* Contraindications to nerve blocks (coagulation defects, infection at puncture site, preexisting neurological deficits in the lower extremities);
* Current severe psychiatric disease or alcoholism or drug dependence;
* Severe visual or auditory disorder;
* Severe complications of DM.

Ages: 65 Years to 90 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: All the participants are more than 65 years with knee osteoarthritis, who will undergo selective total uniknee replacement.Participants(n=150)in diabetes mellitus(DM)group have been diagnosed DM more than three years without severe nervous system complications.participants(n=150)in non diabetes mellitus (NDM)haven't been diagnosed diabetes mellitus.
Sampling Method: Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2013-06; Primary Completion 2014-12 (Estimated); Study Completion 2015-06 (Estimated)

PRIMARY OUTCOMES:
the management of intraoperation | the time during anesthesia and intraoperation

SECONDARY OUTCOMES:
Postoperative recovery by the Post-operative Quality Recovery Scale (PQRS) | 7 days postoperatively
Stress and inflammation | 7 days postoperatively

OTHER OUTCOMES:
postoperative complications | 7 days postoperatively

CONTACTS AND LOCATIONS:
Overall Officials: Zhang Hong, M.D,Ph.D, Study Chair — Professor and Director, Anesthesia and Operation Center, Chinese People's Liberation Army General Hospital
Locations (1):
- Anesthesia and Operation Center, Chinese People's Liberation Army General Hospital, Beijing, Beijing Municipality, China

REFERENCES:
- [Derived] Lu B, Jin J, Pei S, Gong M, Liu J. Anesthesia via peripheral nerve blocks during total knee replacement has no effect on postoperative inflammation in elderly patients. J Orthop Surg (Hong Kong). 2023 Sep-Dec;31(3):10225536231217539. doi: 10.1177/10225536231217539. PMID 38037804
- [Derived] Liu J, Yuan W, Wang X, Royse CF, Gong M, Zhao Y, Zhang H. Peripheral nerve blocks versus general anesthesia for total knee replacement in elderly patients on the postoperative quality of recovery. Clin Interv Aging. 2014 Feb 18;9:341-50. doi: 10.2147/CIA.S56116. eCollection 2014. PMID 24600214